CLINICAL TRIAL: NCT02930421
Title: Clinical and Physiological Effects of Exercise Training in Symptomatic Patients With Mild COPD
Brief Title: Exercise Training in Patients With Mild COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-125; 1141108 (Other: FONDECYT)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: COPD
Keywords: mild COPD; Exercise training; Six minute walking distance; Quality of life; Saint George Respiratory Questionnaire (SGRQ)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (ET) (Experimental): Patients will enter an 8-week ET program of 3 days per week supervised exercise training at the Rehabilitation Physiotherapy Gymnasium. Exercise training will include high-intensity endurance training at 60-80% of baseline peak work rate and strength training of upper and lower limbs with 3 sets of 6 repetitions at 50% of one repetition maximum. Each session will be 60 min duration, 30 min dedicated to cycle exercise.
  Interventions: Other: Exercise training
- Usual care (UC) (No Intervention): The UC group will receive usual outpatient care and follow-up.

INTERVENTIONS:
Other: Exercise training — 30 min of exercise on a cycle ergometer at 80% of HRmax, 30 min of strength training of upper and lower limbs
  Arms: Exercise training (ET)

SUMMARY:
The primary aim of this clinical study is to investigate if exercise training can improve exercise capacity and quality of life in dyspneic mild chronic obstructive pulmonary disease patients.

DETAILED DESCRIPTION:
Peripheral muscle mass and function can be impaired in patients with mild chronic obstructive pulmonary disease (COPD). Quadriceps cross-sectional area is reduced in these patients compared to controls [1], particularly in those with dyspnea as compared to non-dyspneic counterparts and smoker controls [2]. Reduced physical activity is closely related to peripheral muscle mass in mild COPD [1], suggesting that early therapeutic interventions are needed in this group of patients. In addition, reduced quadriceps mass is strongly associated to quadriceps weakness [3,4] and a substantial proportion of patients with mild COPD (28%) had quadriceps weakness [5]. Reduced muscle mass and resultant muscle weakness contribute to limiting exercise in COPD [6-8] and to reduce physical activity, particularly in mild disease [1].

Exercise training (ET) is widely used in patients with moderate-to-very-severe COPD to improve peripheral muscle function and thus exercise capacity and quality of life [9]. Unfortunately, the effects of ET in mild COPD are currently unclear. A recent systematic review identified three low-quality studies with different designs (retrospective, one group pre-posttest, and one randomized controlled trial) [10]. The authors found significant improvements in exercise capacity (effect size 0.87-1.82) and quality of life (effect size 0.24-0.86) after comparing pretest-posttest data and ET with usual care. Although these results are inconclusive and indicate that additional and more robust studies should be conducted [10], current recommendations to initiate ET include even mild disease if dyspnea or exercise limitation are present [11]. Since peripheral muscle mass and function improve with ET [9], the investigators hypothesize that this statement is correct and consequently ET will increase exercise capacity in dyspneic patients with mild COPD in comparison to usual care.

Patients will enter an 8-week ET program of 3 days per week supervised exercise training at the Rehabilitation Physiotherapy Gymnasium. Exercise training will include high-intensity endurance training at 60-80% of baseline peak work rate and strength training of upper and lower limbs with 3 sets of 6 repetitions at 50% of one repetition maximum [12,13]. Each session will be 60 min duration, 30 min dedicated to cycle exercise. The UC group will receive usual outpatient care and follow-up.

The study will require 30 patients per arm to detect an effect size of 0.88 [10] at the 5% significance level and with 80% power, allowing a dropout rate of 30%.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects, aged 45-80 years
* baseline post-bronchodilator forced expiratory volume at one second (FEV1) ≥80% of predicted normal and baseline (post-bronchodilator) FEV1/forced vital capacity (FVC) ≤70%
* current or ex-smokers with a smoking history of at least 10 pack-years
* dyspnea during activities of daily life, defined as modified Medical Research Council (mMRC) scale [0-4 points] ≥1 point

Exclusion Criteria:

* history of asthma or other chronic lung disease (e.g.: interstitial lung disease; sarcoidosis; tuberculosis; cystic fibrosis; bronchiectasis; previous lung resection)
* comorbidities that would prevent the patient from performing an exercise test (including psychological or cognitive disorders): chronic congestive heart failure; recent myocardial infarction [6 months or less]; cardiac arrhythmia requiring drug therapy; neuromuscular and peripheral vascular diseases
* the presence of usual co-morbidities, such as essential hypertension, diabetes, osteoporosis, hypothyroidism, under proper medical control, and obesity, excluding extreme obesity, will not be considered an exclusion criterion.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the six minute walking distance | Baseline and 8 weeks

SECONDARY OUTCOMES:
Change in disease specific quality of life (SGRQ) | Baseline and 8 weeks
  Saint George Respiratory Questionnaire
Change in exercise time during constant-load cycle exercise | Baseline and 8 weeks
  Constant-load exercise at 70% of peak baseline workload

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Díaz, Principal Investigator — Departamento de Enfermedades Respiratorias
Locations (1):
- Respiratory Department; Hospital Clinico Universidad Catolica, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Shrikrishna D, Patel M, Tanner RJ, Seymour JM, Connolly BA, Puthucheary ZA, Walsh SL, Bloch SA, Sidhu PS, Hart N, Kemp PR, Moxham J, Polkey MI, Hopkinson NS. Quadriceps wasting and physical inactivity in patients with COPD. Eur Respir J. 2012 Nov;40(5):1115-22. doi: 10.1183/09031936.00170111. Epub 2012 Feb 23. PMID 22362854
- [Background] Diaz AA, Morales A, Diaz JC, Ramos C, Klaassen J, Saldias F, Aravena C, Diaz R, Lisboa C, Washko GR, Diaz O. CT and physiologic determinants of dyspnea and exercise capacity during the six-minute walk test in mild COPD. Respir Med. 2013 Apr;107(4):570-9. doi: 10.1016/j.rmed.2012.12.011. Epub 2013 Jan 9. PMID 23313036
- [Background] Bernard S, LeBlanc P, Whittom F, Carrier G, Jobin J, Belleau R, Maltais F. Peripheral muscle weakness in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Aug;158(2):629-34. doi: 10.1164/ajrccm.158.2.9711023. PMID 9700144
- [Background] Seymour JM, Ward K, Sidhu PS, Puthucheary Z, Steier J, Jolley CJ, Rafferty G, Polkey MI, Moxham J. Ultrasound measurement of rectus femoris cross-sectional area and the relationship with quadriceps strength in COPD. Thorax. 2009 May;64(5):418-23. doi: 10.1136/thx.2008.103986. Epub 2009 Jan 21. PMID 19158125
- [Background] Seymour JM, Spruit MA, Hopkinson NS, Natanek SA, Man WD, Jackson A, Gosker HR, Schols AM, Moxham J, Polkey MI, Wouters EF. The prevalence of quadriceps weakness in COPD and the relationship with disease severity. Eur Respir J. 2010 Jul;36(1):81-8. doi: 10.1183/09031936.00104909. Epub 2009 Nov 6. PMID 19897554
- [Background] Baarends EM, Schols AM, Mostert R, Wouters EF. Peak exercise response in relation to tissue depletion in patients with chronic obstructive pulmonary disease. Eur Respir J. 1997 Dec;10(12):2807-13. doi: 10.1183/09031936.97.10122807. PMID 9493665
- [Background] Casaburi R. Limitation to exercise tolerance in chronic obstructive pulmonary disease: look to the muscles of ambulation. Am J Respir Crit Care Med. 2003 Aug 15;168(4):409-10. doi: 10.1164/rccm.2305013. No abstract available. PMID 12912729
- [Background] Singer J, Yelin EH, Katz PP, Sanchez G, Iribarren C, Eisner MD, Blanc PD. Respiratory and skeletal muscle strength in chronic obstructive pulmonary disease: impact on exercise capacity and lower extremity function. J Cardiopulm Rehabil Prev. 2011 Mar-Apr;31(2):111-9. doi: 10.1097/HCR.0b013e3182033663. PMID 21240003
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Jacome C, Marques A. Pulmonary rehabilitation for mild COPD: a systematic review. Respir Care. 2014 Apr;59(4):588-94. doi: 10.4187/respcare.02742. Epub 2013 Oct 8. PMID 24106321
- [Background] Rochester CL, Vogiatzis I, Holland AE, Lareau SC, Marciniuk DD, Puhan MA, Spruit MA, Masefield S, Casaburi R, Clini EM, Crouch R, Garcia-Aymerich J, Garvey C, Goldstein RS, Hill K, Morgan M, Nici L, Pitta F, Ries AL, Singh SJ, Troosters T, Wijkstra PJ, Yawn BP, ZuWallack RL; ATS/ERS Task Force on Policy in Pulmonary Rehabilitation. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1373-86. doi: 10.1164/rccm.201510-1966ST. PMID 26623686
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Background] Langer D, Hendriks E, Burtin C, Probst V, van der Schans C, Paterson W, Verhoef-de Wijk M, Straver R, Klaassen M, Troosters T, Decramer M, Ninane V, Delguste P, Muris J, Gosselink R. A clinical practice guideline for physiotherapists treating patients with chronic obstructive pulmonary disease based on a systematic review of available evidence. Clin Rehabil. 2009 May;23(5):445-62. doi: 10.1177/0269215509103507. Epub 2009 Apr 23. PMID 19389745